CLINICAL TRIAL: NCT04351529
Title: Austrian COVID-19 Registry (AGMT_COVID-19)
Brief Title: Austrian COVID-19 Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_COVID-19
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Infectious Disease; COVID-19
MeSH Terms: conditions — Communicable Diseases; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The AGMT_COVID-19 Registry is designed as multicenter observational cohort of patients, that are tested positive for SARS-CoV-2. Data will be collected from all sites in Austria willing to participate.

Due to the non-interventional nature of the AGMT_COVID-19 registry, only routine data, which has already been recorded in the patient's medical chart, is transferred to the eCRF.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The disease was first identified at the end of 2019 in Wuhan, the capital of Hubei province in central China, and has since spread globally.

There are currently no authorised vaccines or treatments in the EU (European Union) to prevent or treat novel coronavirus disease (COVID-19) specifically or any other coronaviruses.

The AGMT_COVID-19 Registry is designed as multicenter observational cohort of patients, that are tested positive for SARS-CoV-2. Data will be collected from all sites in Austria willing to participate.

Due to the non-interventional nature of the AGMT_COVID-19 registry, only routine data, which has already been recorded in the patient's medical chart, is transferred to the eCRF. Treatment indication, the decision to offer treatment, treatment choice, dose, schedule and dose reductions/escalations, and response assessments shall be exclusively based on the risk/benefit estimation of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Positive test for SARS-CoV-2

Exclusion Criteria:

* Due to the non-interventional design of the registry there are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The AGMT_COVID-19 Registry is designed as multicenter observational cohort of patients, that are tested positive for SARS-CoV-2.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Documentation of natural course and the therapeutic landscape of patients with COVID-19. | 2 years
  Due to the non-interventional nature of the AGMT_COVID-19 registry, only routine data, which has already been recorded in the patient's medical chart, is transferred to the eCRF. Treatment indication, the decision to offer treatment, treatment choice, dose, schedule and dose reductions/escalations, and response assessments shall be exclusively based on the risk/benefit estimation of the treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — IIIrd Medical Department, Private Medical University Hospital Salzburg
Locations (4):
- Austria (4):
  - LKH Feldkirch: Innere Medizin II/ Interne E (Hämatologie und Onkologie), Feldkirch
  - Kepler Universitätsklinikum Linz, Med. Campus III., Klinik für Lungenheilkunde / Pneumologie, Linz
  - IIIrd Medical Department, Private Medical University Hospital Salzburg, Salzburg
  - KH Zams: Innere Medizin Internistische Onkologie und Hämatologie, Zams